CLINICAL TRIAL: NCT00759707
Title: Endothelial Function in Lower Extremity Bypass Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua A. Beckman, MD, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2006P-000424
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Arterial Disease
Keywords: saphenous vein bypass grafts; flow-mediated vasodilation
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigators who analyzed the results of vascular function testing were blinded to the participant identity.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): ultrasound imaging of saphenous vein bypass graft following an ischemic stimulus, administration of sublingual nitroglycerin and intravenous administration of L-NMMA.
  Interventions: Drug: L-N^G monomethyl arginine (L-NMMA)

INTERVENTIONS:
Drug: L-N^G monomethyl arginine (L-NMMA) — L-NMMA was infused at a dose of 1 mg/kg over 10 minutes to competitively inhibit the production of nitric oxide. Ultrasound imaging of the saphenous vein [arterial] bypass at baseline, and following an ischemic stimulus, administration of sublingual nitroglycerin, and intravenous administration of L-NMMA.

SUMMARY:
This study will determine whether or not saphenous vein [arterial] bypass grafts in the leg relax in response to increases in blood flow.

DETAILED DESCRIPTION:
Subjects who have undergone saphenous vein [arterial] bypass grafts from the femoral to above-knee popliteal artery will undergo ultrasound imaging at rest, and again after 5 minutes of blood pressure cuff occlusion of the calf. (at 1 minute and 15 minutes) Subjects will then be given sub-lingual nitroglycerin, and repeat ultrasound will be performed 3 minutes later. Following 10 minutes of rest, subjects will be given intravenous L-NMMA, a specific nitric oxide inhibitor, to help determine the responsible agent of the vein graft flow mediated dilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have undergone femoral artery to above-knee popliteal artery saphenous vein bypass grafts

Exclusion Criteria:

* Amputation beyond the toes
* Critical limb ischemia defined as rest pain, non-healing ulceration or gangrene
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Beckman, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population: All 19 study subjects had continuously patent femoral-to-popliteal arterial bypass with autogenous greater saphenous vein. Ultrasound imaging of saphenous vein bypass graft followed an ischemic stimulus and administration of sublingual nitroglycerin. In the last 6 consecutive subjects, L-N^G monomethyl arginine (L-NMMA) was administered intravenously.
Period: Overall Study
Arm/Group | Study Population
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Population
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Saphenous Vein Bypass Graft Vasodilation
Description: Flow-mediated, endothelium-dependent vasodilation was determined by comparing baseline vein graft diameter with vein graft diameter as measured after deflation of a 2.5-inch wide sphygmomanometric cuff that had been inflated to suprasystolic pressure for 5 minutes. The cuff was never placed directly over the graft. Vasodilation of the vein graft was determined by acquiring images at 1 minute after cuff deflation.
Time Frame: Single visit study
Measure: Mean (Standard Error); unit: vein bypass graft size increase (%)
Arm/Group | Study Population
Number analyzed (Participants) | 19
vein bypass graft size increase (%) | 5.28 (3.1)

ADVERSE EVENTS:
Time Frame: 1 month after the study day.
Description: It does not differ.
Groups:
- Study Population: All 19 study subjects. Each subject qualified for the study on the basis of a continuously patent femoral-to-popliteal arterial bypass with autogenous greater saphenous vein.
Arm/Group | Study Population
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No